CLINICAL TRIAL: NCT01097512
Title: A Phase I, Dose-escalation Study of a Combination AS703569 and Gemcitabine Given to Subjects With Advanced Malignancies
Brief Title: AS703569 and Gemcitabine Combination in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27902
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: AS703569; MSC1992371A; Aurora kinase inhibitor; Cancer treatable with gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MSC1992371A; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen 1: AS703569/gemcitabine (Experimental): Gemcitabine on Days 1 and 8, AS703569 on Days 2 and 9, of a 21-day cycle
  Interventions: Drug: AS703569/gemcitabine
- Regimen 2: AS703569/gemcitabine (Experimental): AS703569 on Days 1 and 8, gemcitabine on Days 2 and 9, of a 21-day cycle
  Interventions: Drug: AS703569/gemcitabine

INTERVENTIONS:
Drug: AS703569/gemcitabine — Gemcitabine on Days 1 and 8, AS703569 on Days 2 and 9, of a 21-day cycle. The starting dose (DL1) for AS703569 will be 10mg/m2/day. The subsequent dose levels of AS703569 will follow the dose-escalation scheme with an approximate 50% increase from DL1 to DL2, 40% from DL2 to DL3, and thereafter an approximate increase of 33% from one dose level to the next.
  Gemcitabine will be administered at the dose of 1000mg/m2 once weekly during the first two weeks of each 21-day cycle.
  Other Names: Aurora kinase inhibitor; MSC1992371A
  Arms: Regimen 1: AS703569/gemcitabine
Drug: AS703569/gemcitabine — AS703569 on Days 1 and 8, gemcitabine on Days 2 and 9, of a 21-day cycle. The starting dose (DL1) for AS703569 will be 10mg/m2/day. The subsequent dose levels of AS703569 will follow the dose-escalation scheme with an approximate 50% increase from DL1 to DL2, 40% from DL2 to DL3, and thereafter an approximate increase of 33% from one dose level to the next.
  Gemcitabine will be administered at the dose of 1000mg/m2 once weekly during the first two weeks of each 21-day cycle.
  Other Names: Aurora kinase inhibitor; MSC1992371A
  Arms: Regimen 2: AS703569/gemcitabine

SUMMARY:
In clinical practice and research, combination of anticancer agents is often used to improve efficacy of treatment. In vitro and in vivo experiments have shown additive-synergistic anti-tumour effects of AS703569 treatment when combined with gemcitabine. Specifically, additive-synergistic anti-tumour effects were noticed when the two agents were given sequentially and not concomitantly i.e. AS703569 given the day before or the day after gemcitabine. This trial was designed to investigate in parallel two regimens testing sequential administration of AS703569 either the day after gemcitabine infusion, (Regimen 1) or the day before (Regimen 2).

ELIGIBILITY:
Inclusion Criteria:

Histologically/cytologically confirmed diagnosis of measurable or assessable malignancy, who meets one of the following conditions:

Subject with a tumour for which gemcitabine is approved, Subject with a tumour for which gemcitabine is considered standard of care, Subject with other tumour type either refractory or intolerant to or for whom there is not an accepted standard treatment.

Male or female with at least 18 years of age. Life expectancy of at least 3 months.

Eastern Cooperative Oncology Group (ECOG) Performance Status < 2.

No more than 3 prior chemotherapy regimens for advanced/metastatic disease.

At least 4 weeks since last chemotherapy, hormonal therapy, immunotherapy, biological or any other pharmacological or investigational treatment or radiotherapy (6 weeks wash-out for nitrosoureas and mitomycin C, 5 half-lives for non-cytotoxics). Subjects on chronic hormonal therapy may continue with the same treatment unchanged.

Adequate renal, hepatic and bone marrow functions (assessed 7 days before inclusion in the trial) as defined by:

Serum creatinine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 21 days
  To determine the maximum tolerated dose (MTD) during a 21-day cycle, for each of the two planned regimens using combination therapy with AS703569 and gemcitabine.

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAE) | Minimum 21 days or 1 cycle
  Proportion/number of subjects with TEAE's during the first and subsequent treatment cycles in each cohort for each of the 2 regimens.
Progression-Free Survival (PFS) time (For subjects with locally advanced /metastatic pancreatic cancer included after completion of the dose escalation part) | Variable
  PFS time is defined as time (in months) from first drug intake to date of progression as reported and documented by the investigator (i.e. radiological progression per Response Evaluation Criteria in Solid Tumors [RECIST] criteria) or death from any cause.
Time to Tumor Progression (TTP) time (For subjects with locally advanced /metastatic pancreatic cancer included after completion of the dose escalation part) | Variable
  TTP time is defined as the time (in months)from first drug intake to the date of progression, as reported and documented by the Investigator (i.e. radiological progression per RECIST).
Overall Survival (OS) time (For subjects with locally advanced /metastatic pancreatic cancer included after completion of the dose escalation part) | Variable
  OS time is defined as the time (in months) from first drug intake to any cause of death.
Progressive disease (PD) | Every other cycle
  Proportion of patients with progressive disease as assessed at the end of every other cycle according to disease-specific guidelines
Best overall response (For subjects with locally advanced /metastatic pancreatic cancer included after completion of the dose escalation part) | Every other cycle
  For subjects with locally advanced /metastatic pancreatic cancer:
  Best overall response: presence of at least one confirmed Complete Response (CR) or confirmed Partial Response (PR) (using RECIST v1.0) during treatment in the 2 regimens as assessed at the end of every other cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Narmyn Rejeb, MD, Study Director — Merck Serono S.A., Geneva
Locations (3):
- Institut Jules Bordet, Brussels, Belgium
- France (2):
  - Service Inter-Hospitalier de Canderologie Bichat-Beaujon (SIHC) Hopital Beaujon, Clichy
  - Unite d'Oncologie Medicale Hopital COCHIN, Paris

REFERENCES:
- [Result] Raymond E, Alexandre J, Faivre S, Goldwasser F, Besse-Hammer T, Gianella-Borradori A, Jego V, Trandafir L, Rejeb N, Awada A. A phase I schedule dependency study of the aurora kinase inhibitor MSC1992371A in combination with gemcitabine in patients with solid tumors. Invest New Drugs. 2014 Feb;32(1):94-103. doi: 10.1007/s10637-013-9950-y. Epub 2013 Mar 29. PMID 23539344